CLINICAL TRIAL: NCT07316543
Title: Cognitive and Functional Telehealth-based Assessment and Intervention in Veterans With Psychogenic Nonepileptic Seizures
Brief Title: Cognitive Rehabilitation for Veterans With PNES
Acronym: CRVWP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRD9-001-25M; 1IK2RD000605-01A2 (Other Grant/Funding Number: VA RRD&T)
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Psychogenic Nonepileptic Seizures (PNES)
Keywords: functional neurological disorder; functional/dissociative seizures; functional cognitive disorder; cognitive rehabilitation
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Conversion Disorder | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Development of a cognitive rehabilitation intervention to improve cognition and everyday functioning for Veterans with PNES.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): Single arm of pilot trial testing the cognitive rehabilitation intervention
  Interventions: Behavioral: Cognitive Rehabilitation And Functional Treatment (CRAFT)

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation And Functional Treatment (CRAFT) — Cognitive rehabilitation tailored to improve cognition and participation in daily activities for Veterans with PNES

SUMMARY:
Psychogenic nonepileptic seizures (PNES) reflect a subtype of functional neurological disorder (FND) that is common and extremely disabling in Veterans. Cognitive problems are highly prevalent in PNES, they reduce quality of life, and they severely limit daily functioning. Currently, there are no available treatments that target cognition to improve daily function in PNES or other FNDs, leaving a major gap in the literature. Cognitive re-habilitation improves daily functioning in Veterans with related neuropsychiatric disorders and has a high chance of success in Veterans with PNES. The proposed study will solicit direct input from Veterans with PNES via qualitative interviews to inform the design of a cognitive treatment workbook. The workbook will then be iteratively refined based on participatory feedback from Veterans with PNES and their treatment providers. The full cognitive intervention protocol will be pilot tested to inform a fully powered RCT. Results will support a line of research that aims to improve cognition and function in Veterans with PNES and related FNDs.

DETAILED DESCRIPTION:
Significance to VA: A cognitive intervention for Veterans with psychogenic nonepileptic seizures (PNES) and other functional neurological disorders (FNDs) is desperately needed. FNDs such as PNES are prevalent, underrecognized, and highly disabling in Veterans. Cognitive dysfunction is one of the most common and disabling symptoms in PNES and other FNDs, it contributes to reduced quality of life, and it is not adequately ad-dressed by available treatments. RCTs examining cognitive rehabilitation interventions in related disorders (e.g., TBI) have repeatedly shown that improving cognition leads to improvements in everyday functioning, including work, school, medication management, and driving. Therefore, a similar approach to treating cognitive problems in Veterans with PNES is very likely to improve their everyday functioning. The current CDA2 project will develop and pilot test a cognitive intervention, adapted from prior successful treatments (e.g., in TBI), and tailored to Veterans with PNES. Because of strong overlap between PNES and other FNDs, the intervention from this CDA2 will be ideally suited for adaptation for the >60,000 U.S. Veterans with any subtype of FND.

Innovation and Impact: This is the first study to develop and pilot test an intervention, grounded in a rehabilitation framework and Veteran participant feedback, to improve cognition and daily functioning in Veterans with PNES. Telehealth will be used for all aspects of the current project, facilitating nationwide study recruitment. Telehealth will improve representativeness of the current study sample (enhancing generalizability) and will increase Veteran access to the intervention by reducing barriers to treatment. Strategies from implementation science (e.g., participatory Veteran research) will be infused into the intervention from the start. This will lead to a cognitive intervention that is ideally suited for dissemination and sustainability in VA clinics nationwide.

Specific Aims:

Aim 1: Explore the impact of cognition on daily function via qualitative interviews in 15 Veterans with PNES.

H1: Problems in attention/processing speed will be related to worse daily function in Veterans with PNES.

Aim 2: Develop a feasible telehealth-based cognitive rehabilitation workbook for improving daily functioning in Veterans with PNES, informed by feedback from 12 Veterans with PNES and 12 treatment providers.

H2: The cognitive workbook for improving everyday functions will show promise, as measured by mean workbook ratings of 4 on the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) in Veterans with PNES and PNES treatment providers.

Aim 3: Evaluate feasibility of the cognitive treatment with a pilot single arm trial in 20 Veterans with PNES.

H3a: Veterans with PNES will rate the cognitive treatment protocol, including functional outcome measures, as acceptable, appropriate, and feasible, based on mean ratings of 4 on the AIM, IAM, and FIM, respectively.

H3b: Veterans with PNES will show improvement in the co-primary outcomes of cognition and daily functioning, with at least a small to moderate effect size (d 0.30).

Methodology: Veterans with PNES will be recruited from 19 nationwide VA Epilepsy Centers of Excellence sites. Feasibility of recruitment is supported by my VISN1 CDA study. CDA2 Study 1 will analyze qualitative interview data in Veterans with PNES to inform workbook development. Study 2 will develop a cognitive treatment workbook, with the AIM, IAM, and FIM as outcomes. Study 3 will pilot test the intervention, with feasibility (AIM, IAM, and FIM), and composite cognition and daily function (WHODAS 2.0) scores as outcomes.

Path to Translation/Implementation: This CDA2 responds to a golden opportunity to develop, refine, and pilot test a workbook-based cognitive intervention for Veterans with PNES. The cognitive intervention will be well suited for a subsequent fully powered RCT (an anticipated VA Merit Award), which can demonstrate efficacy and effectiveness. Because the cognitive intervention will be designed with implementation in mind from the start, it will be perfectly positioned for immediate dissemination and sustainability within the VA system.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran
* able to provide informed consent
* reports cognitive difficulties
* prior video EEG diagnosis of PNES
* English speaking
* able to read at least at 8th grade level
* access to a private space with a computer (13-inch monitor)
* internet access

Exclusion Criteria:

* acute psychosis (hallucinations or delusions)
* current active suicidality
* a diagnosis of dementia or intellectual disability
* sensory impairment (e.g., deafness) that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
WHODAS 2.0 Total Score | Once at baseline (prior to the intervention) and once following the 8-12 week intervention.
  Everyday functioning as measured by the World Health Organization Disability Assessment Schedule 2.0, range = 0-100, higher scores = greater disability.

SECONDARY OUTCOMES:
Cognitive Composite | Once at baseline (prior to the intervention) and once following the 8-12 week intervention.
  Composite of scores from standardized neuropsychological tests measuring multiple cognitive domains. Because this measure is a composite of many individual cognitive test scores, it will be represented by a Z-score and does not have a minimum or maximum value.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan A Van Patten, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
One or more data sets without personal identifiers will be generated during the data analysis phase of this study. The data sets will include all data underlying any publications generated by this study and therefore these will be sufficient to reproduce or verify any published findings. The final data set(s) for this study will be maintained locally at VA Providence until enterprise-level resources become available for long-term storage and access.
Supporting Information: Study Protocol, SAP, Analytic Code